CLINICAL TRIAL: NCT00160511
Title: A Double-blind, Randomized, Placebo-controlled, Parallel-group, 16 Week, Multicenter Trial Evaluating the Efficacy and Safety of Levetiracetam 500 mg Tablets in Bid Administration (Daily Dose Ranging From 1000 mg to 3000 mg), in Adults (≥ 18 Years of Age) Suffering From Postherpetic Neuralgia
Brief Title: A 16 Week Study Evaluating Levetiracetam in the Treatment of Post Herpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01087
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-09

CONDITIONS: Neuralgia, Postherpetic
Keywords: Postherpetic Neuralgia (PHN); Levetiracetam; Keppra; Nerve Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
16 week trial assessing the efficacy, safety, and tolerability of levetiracetam compared with placebo in the treatment of postherpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* male or female outpatient greater than or equal to 18 years of age.
* suffering presently from neuralgia, which has been present for at least 3 months since healing of acute herpes zoster skin rash.
* PHN pain at entry into the study must meet the following criteria: a VAS of at least 40 mm at visit 2 (to assess pain intensity during the past week) and with an average daily score of at least 4 on the PIS during the baseline period as evaluated on a minimum of 4 days.
* an estimated creatinine clearance of at least 50 ml/min.

Exclusion Criteria:

* receiving professional psychological support (such as cognitive behavioral therapy) currently or within 2 weeks prior to visit 1 specifically for coping with PHN.
* previous neurolytic or neurosurgical therapy for PHN, at any time in the subject's history or treatment with TENS (transelectroneuro stimulation) currently or within the past 2 weeks.
* known co-existent source of pain or painful peripheral neuropathy.
* known significant neurological disorder other than the study disease or a condition which can mimic stroke with distal neurological deficit (amyotrophy, radiculopathy, history of TIAs, multiple sclerosis, or any amputations).
* conditions known to be associated with immunosuppressive states.
* clinically significant major depression defined as a Beck Depression Inventory Score > 21 at selection including those with a history of Bipolar Disorder.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 2004-04; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of levetiracetam in the treatment of Post Herpetic Neuralgia by measuring the absolute change in the average weekly Pain Intensity Scale (PIS).

SECONDARY OUTCOMES:
Assess the efficacy, safety and tolerability of levetiracetam in the treatment of Post Herpetic Neuralgia; Reduction in the mean PIS over the last week of the evaluation period compared to the baseline period.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma